CLINICAL TRIAL: NCT01564394
Title: Effects of Qigong on Fatigue & Quality of Life in Elderly Prostate Cancer Survivors
Brief Title: Body Mind Training Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Anita Kinney, Jon & Karen Huntsman Presidential Professor in Cancer Research, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: U of Utah COA Pilot Grant
Record Dates: First submitted 2012-03-22; First posted 2012-03-27 (Estimated); Results first posted 2015-08-19 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-11

CONDITIONS: Cancer Related Fatigue
Keywords: qigong; mindfulness meditation; fatigue; prostate cancer
MeSH Terms: conditions — Fatigue; Prostatic Neoplasms | interventions — Qigong

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Qigong (Experimental): Qigong originated in China hundreds of years ago and has been practiced for centuries. It consists of a sequence of slow, flowing physical movements with concentration on the breath and awareness and may promote physical and mental relaxation and energy balance.
  Interventions: Behavioral: Qigong
- Stretching control (Sham Comparator): The non-aerobic stretching will serve as an attention control group to control for non-specific factors; dose of attention and to mimic being in a group setting.
  Interventions: Behavioral: Non-aerobic stretching

INTERVENTIONS:
Behavioral: Qigong — Classes will be 60 minutes in duration, held two times a week, supplemented with home-based sessions over 12 weeks. The classes will be led by a trained Qigong instructor and consist of postures, movements, deep breathing techniques and meditation. It will include eccentrically-biased Qigong movements with an emphasis on weight shifting and posture control. The continuous body movements coupled with progressively diminishing base of support, dynamic challenge to balance, and concentration on body positions requiring eccentric muscle activity should improve the levels of fatigue and quality of life in older prostate cancer survivors.
  Arms: Qigong
Behavioral: Non-aerobic stretching — The non-aerobic stretching classes will serve as an attention control. They will be 60 minutes in duration, held two times a week, supplemented with home-based sessions over 12 weeks. They will be led by an Huntsman Cancer Institute (HCI) fitness specialist and will consist of light stretching exercises; while avoiding a focus on meditation.
  Arms: Stretching control

SUMMARY:
Aim 1: Assess the feasibility, safety and efficacy of a Qigong intervention in elderly prostate cancer survivors.

Describe participation, retention, and adherence rates and assess reasons for participation, attrition, and non-adherence.

Identify effective recruitment and retention strategies. Ascertain participants' level of satisfaction and additional perceptions of the experimental and control interventions, perceived study burden, study design, and implementation.

Aim 2: Provide preliminary data on potential effects of Qigong vs. non-aerobic stretching exercises on fatigue, psychosocial outcomes, and health-related quality of life in preparation for a future R01 application for a larger, definitive randomized controlled trial. Hypothesis: Qigong participants will have improved fatigue levels, quality of life, and related psychosocial and health outcomes compared to those randomized to the non-aerobic stretching group.

DETAILED DESCRIPTION:
This ongoing feasibility study is a two-armed, parallel group, randomized clinical trial.We will recruit 60 elderly prostate cancer survivors (age 55+ years) and their significant others (spouse, domestic partner, or close family member).

Considering literature attesting to strains associated with caregiver status, we will also collect survey and physical assessment data to explore the intervention's effect on significant others.

Recruitment occurs through Huntsman Cancer Institute's outpatient clinic and University and community-based strategies (for example, newspaper ads, flyers, support groups, patient registries).

We will measure relevant psychosocial measures, including fatigue and quality of life (SF36 & EPIC), perceived stress, distress, mood, cognitive function, social connectedness, demographics, and leisure time, at baseline, the six-week midpoint, and one week post-intervention. Weekly measures of fatigue and quality of life and physical activity logs will also be administered.

Biometric assessments, including balance and mobility, flexibility, blood pressure, resting heart rate, body mass index, and waist-hip-ratio, will be done at baseline (before randomization) and one week post-intervention.

Significant others will undergo the same survey measures as the prostate cancer survivors, except for measures specific to prostate cancer (e.g., EPIC-26-short form).

Participants will be recruited in two cohorts, one beginning early March and the other early June, 2012. The twice-weekly exercise classes will be 60 minutes in duration, running for 12 weeks. Classes will be conducted at Huntsman Cancer Institute's Survivor & Wellness Center, beginning one week after baseline physical assessments. Participants will receive a DVD of the respective class led by trained and qualified instructors so they can supplement classes with home-based sessions.

Qigong class will consist of postures, movements, deep breathing techniques, and meditation, including an emphasis on weight shifting, breath, and posture control.

Non-aerobic stretching will consist of light stretching exercises that avoid focus on meditation. This class will serve as the control group for non-specific factors such as attention dose and the group setting.

To ensure consistency of physical intensity between the two study arms, both objective (heart rate monitors) and subjective (self-reported ten-point Borg scale) measures will be performed on participants.

ELIGIBILITY:
Inclusion Criteria:

* Significant fatigue as assessed during screening with the NCI Common Terminology Criteria for Adverse Events (CTCAE) Safety Profiler of fatigue using a cut-off value of ≥ 1; and/or with a fatigue grading scale (general questions that assess level of fatigue currently and in the past week from a scale of 0-100) with a cut off value of >20
* Are sedentary as defined by <150 minutes of mild, moderate, or intense intensity exercise/week per Centers for Disease Control and Prevention(CDC) guidelines
* Able to speak and read English fluently, and understand informed consent
* Reside within 60 miles of Huntsman Cancer Institute and have access to regular transportation to all assessments and intervention classes at HCI
* Willing to: sign a medical record release form; be randomized and willing to participate in classes and all baseline and follow-up appointments
* Significant others and domestic partners of elderly prostate cancer survivors will be eligible if they are at least 18 years of age, read and speak English, willing to sign an informed consent, and provide a physician's release for exercise

Exclusion Criteria:

* Clinical evidence of metastatic disease other than elevated prostate-antigen specific (PSA) levels
* Current practice of Qigong, Tai Chi or other similar types of Complementary and Alternative medicine that may share similar principles of Qigong
* Inability to pass the Folstein Mini Mental Status Exam (score <23)
* Unable to drive or secure transportation to complete all aspects of the study
* Health conditions (e.g. severe hearing loss, respiratory, cardiovascular, or neurological problems) that might interfere with the required intervention
* Unwilling to be randomized to study groups and/or commit to 12 weeks of Qigong or non-aerobic stretching classes

Ages: 55 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anita Kinney, RN, PhD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (2):
- United States (2):
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 502 senior prostate cancer survivors in Utah through clinic referrals, registries, community advertisements, and community-based support groups.
Pre-assignment Details: Out of 89 prostate cancer survivors screened for eligibility, forty were eligible and interested in participating in the study.Twenty family members met criteria for participating. Only the survivors were randomized to study arms. Family members attended the study arm that the survivor was randomized to.
Groups:
- Qigong: Qigong originated in China hundreds of years ago and has been practiced for centuries. It consists of a sequence of slow, flowing physical movements with concentration on the breath and awareness and may promote physical and mental relaxation and energy balance.
  Qigong : Classes will be 60 minutes in duration, held two times a week, supplemented with home-based sessions over 12 weeks. The classes will be led by a trained Qigong instructor and consist of postures, movements, deep breathing techniques and meditation. It will include eccentrically-biased Qigong movements with an emphasis on weight shifting and posture control. The continuous body movements coupled with progressively diminishing base of support, dynamic challenge to balance, and concentration on body positions requiring eccentric muscle activity should improve the levels of fatigue and quality of life in older prostate cancer survivors.
- Stretching Control: The non-aerobic stretching will serve as an attention control group to control for non-specific factors; dose of attention and to mimic being in a group setting.
  Non-aerobic stretching : The non-aerobic stretching classes will serve as an attention control. They will be 60 minutes in duration, held two times a week, supplemented with home-based sessions over 12 weeks. They will be led by an Huntsman Cancer Institute (HCI) fitness specialist and will consist of light stretching exercises; while avoiding a focus on meditation.
Period: Overall Study
Arm/Group | Qigong | Stretching Control
Started | 30 (Prostate cancer survivors n=20, family n=10. Only survivors were randomized.) | 30 (Prostate cancer survivors n=20, family n=10. Only survivors were randomized.)
Completed | 24 (Prostate cancer survivors n=16, family n=8.) | 20 (Prostate cancer survivors n=13, family n=7.)
Not Completed | 6 | 10
Not completed — Withdrawal by Subject | 6 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Qigong | Stretching Control | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 16
  >=65 years | 23 | 21 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (9.6) | 71.2 (10.1) | 71.2 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 20 | 21 | 41
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Secondary Outcome: Brief Symptom Inventory (BSI)-18 Change From Baseline to 13-weeks
Description: The BSI-18 assesses global distress and three subscales (anxiety, depression, & somatization). Scores are converted to T-scores based on US population norms. Negative change scores indicate improvement in distress. We report data separately for prostate cancer survivors and family members. Based on the population norm a T-score of 63 or above indicates heightened global distress.
Time Frame: Baseline to 13-weeks
Population: Data is presented for Qigong participants (n=16) and family members (n=8 ) and for Stretching participants (n=13) and family members (n=7) .
Measure: Median (Inter-Quartile Range); unit: T-Score
Arm/Group | Qigong | Stretching Control
Number analyzed (Participants) | 24 | 20
T-Score
  Prostate Cancer Survivors Global Index Change | -7.0 [-12.0 to -3.2] | 0.0 [-4.0 to 1.5]
  Prostate Cancer Survivors Anxiety Change | -7.5 [-8.0 to 0.0] | 0.0 [0.0 to 7.5]
  Prostate Cancer Survivors Somatization Change | -6.5 [-10.7 to -0.2] | 0.0 [-4.0 to 2.0]
  Prostate Cancer Survivors Depression Change | -6.5 [-12.0 to 0.0] | 0.0 [-6.5 to 0.5]
  Family Member Global Index Change | -3.5 [-7.7 to 0.0] | -2.0 [-13.0 to 3.0]
  Family Member Anxiety Change | -1.0 [-3.7 to 0.0] | -7.0 [-8.0 to 0.0]
  Family Member Somatization Change | 0.0 [-6.7 to 0.0] | 0.0 [-6.0 to 7.0]
  Family Member Depression Change | -5.0 [-6.7 to 0.0] | -3.0 [-10.0 to 0.0]

2. Primary Outcome: Retention Rate in Study (Feasibility Outcome)
Description: The retention rate was the proportion of participants who remained enrolled in the study and completed post-intervention measures. Range of retention rate is 0 to 1. Prostate cancer survivors were the population targeted in this intervention, therefore, the retention and attendance rates only include prostate cancer survivors (i.e., family members were not included in these calculations).
Time Frame: 13-weeks
Measure: Number; unit: proportion of participants
Arm/Group | Qigong | Stretching Control
Number analyzed (Participants) | 20 | 20
proportion of participants | 0.80 | 0.65

3. Primary Outcome: Attendance Rates in Study (Feasibility Outcome)
Description: The class attendance rates were the number of classes attended by participants divided by the total number of classes offered. Range of attendance rate is 0 to 1. Prostate cancer survivors were the population targeted in this intervention, therefore, the retention and attendance rates only include prostate cancer survivors (i.e., family members were not included in these calculations).
Time Frame: 13-weeks
Measure: Number; unit: Proportion of classes
Arm/Group | Qigong | Stretching Control
Number analyzed (Participants) | 20 | 20
Proportion of classes | 0.85 | 0.68

4. Primary Outcome: FACIT-Fatigue Change From Baseline to 13-weeks.
Description: Our primary outcome of change in fatigue was assessed with the Functional Assessment Chronic Illness Therapy (FACIT)-Fatigue scale. This 13-item scale assesses levels of fatigue during daily activities over the past seven days. Higher scores indicate less fatigue (score range = 0 - 52). Positive change scores indicate improved fatigue.
Time Frame: Baseline to 13-weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Units on scale
Arm/Group | Qigong | Stretching Control
Number analyzed (Participants) | 24 | 20
Units on scale
  Prostate Cancer Survivor FACIT-Fatigue Change | 5.0 [2.0 to 12.7] | 0.0 [-5.5 to 4.5]
  Family Member FACIT-Fatigue Change | 2.5 [-0.7 to 6.0] | 0.0 [-2.0 to 5.0]

ADVERSE EVENTS:
Arm/Group | Qigong | Stretching Control
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No